CLINICAL TRIAL: NCT02217514
Title: Effects of 100 mg and 500 mg BI 44370 TA Orally Applied as 50 mg Tablets on the Pharmacokinetics of 2 mg Orally Administered Midazolam Solution. An Open-label, Randomised, Parallel Group, Fixed-sequence Study With Intraindividual Comparison of Midazolam Pharmacokinetics With and Without BI 44370 TA
Brief Title: Effects of BI 44370 TA Orally Applied as Tablets on the Pharmacokinetics of Orally Administered Midazolam Solution in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1246.3
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

ARMS (5):
- Treatment sequence 1 in male subjects (Experimental): Midazolam alone and 1 h after low dose BI44370BS in male subjects
  Interventions: Drug: Midazolam; Drug: BI 44370 low dose
- Treatment sequence 1 in female subjects (Experimental): Midazolam alone and 1 h after low dose BI44370BS followed by medium dose BI 44370 in an additional visit in female subjects
  Interventions: Drug: Midazolam; Drug: BI 44370 low dose; Drug: BI 44370 medium dose
- Treatment sequence 2 (Experimental): Midazolam before and 48 h after high dose BI44370BS
  Interventions: Drug: Midazolam; Drug: BI 44370 high dose
- Treatment sequence 3 (Experimental): Midazolam before and 24 h after high dose BI44370BS
  Interventions: Drug: Midazolam; Drug: BI 44370 high dose
- Treatment sequence 4 (Experimental): Midazolam before and 1 h after high dose BI44370BS
  Interventions: Drug: Midazolam; Drug: BI 44370 high dose

INTERVENTIONS:
Drug: Midazolam
  Other Names: Dormicum®
Drug: BI 44370 low dose
  Arms: Treatment sequence 1 in female subjects; Treatment sequence 1 in male subjects
Drug: BI 44370 medium dose
  Arms: Treatment sequence 1 in female subjects
Drug: BI 44370 high dose
  Arms: Treatment sequence 2; Treatment sequence 3; Treatment sequence 4

SUMMARY:
Evaluation of the long-term (48 h) and short-term (1 h) effects of BI 44370 BS on the pharmacokinetics of midazolam as marker of a possible inhibition of CYP 3A4; safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
* Age ≥21 and Age ≤50 years
* BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good clinical practice (GCP) and the local legislation.

Exclusion Criteria:

* Any finding of the medical examination (including Blood Pressure (BP), Pulse Rate (PR) and Electrocardiogram (ECG)) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 30 days prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >470 ms);
* A history of additional risk factors for Torsade de Pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

For Male Subjects:

* Not willing to use adequate contraception (condom use plus another form of contraception e.g. spermicide, oral contraceptive taken by female partner, sterilisation, intrauterine device (IUD)) during the whole study period from the time of the first intake of study drug until three months after the last intake

For Female Subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception (adequate contraception e.g. sterilisation, intrauterine pessary (IUP), oral contraceptives)
* Inability to maintain this adequate contraception during the whole study period during the whole study period from the time of the first intake of study drug until one month after the last intake

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum concentration of midazolam in plasma) | up to 24 hours after drug administration
AUC0-tz (area under the concentration-time curve of midazolam in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 24 hours after drug administration
AUC0-infinity (area under the concentration-time curve of midazolam in plasma over the time interval from 0 extrapolated to infinity) | up to 24 hours after drug administration

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | Up to 48 hours after drug administration
tmax (time from dosing to maximum measured concentration) | up to 48 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 48 hours after drug administration
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | up to 48 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 48 hours after drug administration
AUCt1-t2 (Area under the concentration-time curve of the analyte in plasma over the time interval t1 to t2) | up to 48 hours after drug administration
λz (terminal rate constant in plasma) | up to 48 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 48 hours after drug administration
MRTp.o. (mean residence time of the analyte in the body after oral administration) | up to 48 hours after drug administration
CL/F (total/apparent clearance of the analyte in plasma after extravascular administration) | up to 48 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 48 hours after drug administration
ratio of AUC0-∞ 1-OH-midazolam / AUC0-∞ midazolam | up to 48 hours after drug administration
Aet1-t2 (amount of BI 44370 BS eliminated in urine from the time point t1 to time point t2) | up to 24 hours after drug administration
fet1-t2 (fraction of BI 44370 BS eliminated in urine from time point t1 to time point t2) | up to 24 hours after drug administration
CLR,t1-t2 (renal clearance of BI 44370 BS from the time point t1 until the time point t2) | up to 24 hours after drug administration
Number of patients with adverse events | up to 8 days after last drug administration
Assessment of tolerability by investigator on a 4-point scale | up to 8 days after last drug administration